CLINICAL TRIAL: NCT00488878
Title: Data Collection for Patients With Low Grade Ovarian Carcinoma
Brief Title: Data Collection for Patients With Low Grade Ovarian or Peritoneal Tumors
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0137; NCI-2020-13341 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2006-0137 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Low Grade Ovarian Serous Adenocarcinoma; Malignant Ovarian Neoplasm; Ovarian Carcinoma; Primary Peritoneal Carcinoma; Primary Peritoneal Low Grade Serous Adenocarcinoma; Psammocarcinoma
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (electronic health record review): Patients' medical records are reviewed for retrospective and prospective data collection. Patients may also have residual tissue samples collected and stored.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Patients' residual tissue samples are collected
Other: Electronic Health Record Review — Medical records are reviewed

SUMMARY:
This study collects information to maintain a database on patients with low-grade ovarian or peritoneal tumors. Collecting information about the type of cancer and treatment, as well as details about follow-up care, may help researchers learn and better understand these tumor types and help develop better treatments for them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To collect, both prospectively and retrospectively, data on disease characterization, treatment, and outcomes for approximately 1600 female patients with low-grade ovarian and peritoneal tumors.

II. To organize clinical information in order to support multifaceted queries of patient characteristics, treatment, and disease outcome data and to facilitate correlation of these characteristics with patient outcome.

III. To have a single data repository, kept on a secure platform that will integrate clinical information and research findings and serve as a secure archive for future research.

SECONDARY OBJECTIVE:

I. To obtain and store human tumor samples in the form of blocks or slides for the purpose of establishing a tumor bank.

OUTLINE:

Patients' medical records are reviewed for retrospective and prospective data collection. Patients may also have residual tissue samples collected and stored.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose disease progressed to a higher-grade carcinoma since the time of original diagnosis:

  * Ovarian tumor of low malignant potential
  * Low-grade serous carcinoma of the ovary
  * Primary peritoneal tumor of low malignant potential
  * Low-grade serous carcinoma of the peritoneum
  * Psammocarcinoma

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a low-grade tumor of Mullerian origin who sought treatment or a second opinion at MD Anderson Cancer Center (MDACC) at any point in the course of their disease and treatment (beginning in January 1950), and patients currently being treated at MDACC or seeking treatment or a second opinion in the future
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2006-05-19 (Actual); Primary Completion 2034-05-01 (Estimated); Study Completion 2035-05-01 (Estimated)

PRIMARY OUTCOMES:
Prospective and retrospective data collection on disease characterization, treatment, and outcomes | Up to 28 years
Organization of clinical information | Up to 28 years
  Will be done in order to support multifaceted queries of patient characteristics, treatment, and disease outcome data and to facilitate correlation of these characteristics with patient outcome.
Creation of a single data repository to integrate clinical information and research findings | Up to 28 years

SECONDARY OUTCOMES:
Collection and storage of human tumor samples for the establishment of a tumor bank | Up to 28 years

CONTACTS AND LOCATIONS:
Overall Officials: David M Gershenson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org